CLINICAL TRIAL: NCT02643056
Title: Phase II Study to Investigate the Efficacy of Panitumumab in Platinum-resistant Advanced Head and Neck Squamous Cance
Brief Title: Study to Investigate the Efficacy of Panitumumab in Platinum-resistant Advanced Head and Neck Squamous Cancer
Acronym: S10PANI01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southern Europe New Drug Organization (Other)
Collaborators: Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Principal Investigator, Tatiana Terrot, Project Manager, Oncology Institute of Southern Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S10PANI01
Record Dates: First submitted 2015-12-08; First posted 2015-12-30 (Estimated); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Advanced Head and Neck Squamous Cancer
MeSH Terms: interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab (Experimental): 6 mg/kg per administration
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — IV administration every 2 weeks

SUMMARY:
Phase II, multicenter, open labelled, uncontrolled study to evaluate the efficacy and safety profile of panitumumab in patients affected by Head and Neck cancer after at least one cisplatin or carboplatin-based chemotherapy. A translational research study is also planned to evaluate Estimated Glomerular Filtration Rate (EGFR) status by FISH, KRAS, B-RAF, HRAS, NRAS and PIK3CA mutation by DNA sequencing, PTEN protein expression by immunohistochemistry, and Human Papilloma Virus (HPV) genotyping by reverse hybridization.

Panitumumab is administered iv on days 1 and 15 of a 28 days cycle, until progressive disease, unacceptable toxicity, pregnancy, or patient's refusal

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2, not pregnant.
* Histologically or cytologically confirmed Squamous Cell Cancer of the Head and Neck either metastatic or recurrent, judged incurable by surgery or radiation.
* Baseline tumor tissue, sufficient material available for EGFR determination (therapeutic target of panitumumab) and biomarker studies. Patients without available tissue at baseline or with tissue collected longer than 1 year before, may undergo tumor biopsy.
* Progression after or not responding to treatment with at least one cis-platin or carboplatin containing regimen.
* Measurable disease (Response Evaluation Criteria in Solid Tumours - RECIST 1.1).
* Adequate hematological values, renal and hepatic function.
* Patients may not be receiving any other investigational agents

Exclusion Criteria:

* Platinum-naïve patients.
* Patients previously progressed after a regimen containing EGFR-inhibiting agents (as cetuximab, panitumumab, gefitinib, erlotinib), even if there was an initial response.
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) 1 year before enrollment/randomization.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest computed tomography scan.
* Known or suspected brain metastases.
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent
* Known hypersensitivity to panitumumab active ingredient or excipients.
* Any concomitant drugs contraindicated for use with the trial drug according to the Swissmedic approved product information - Human Immunodeficiency Virus (HIV) positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Rate of tumor response in advanced platinum-resistant head and neck cancer | Radiological tumor evaluation every 8 weeks, minimum 12 weeks
  To evaluate rate of radiological tumor response in advanced platinum-resistant head and neck cancer

SECONDARY OUTCOMES:
Adverse Event according to Common Terminology Criteria for Adverse Events (CTCAE) v.3 | Collection of adverse event for at least the first 8 weeks
  To collect all adverse event occurred during the treatment
Analysis of tumor biomarkers | 28 days (1 cycle)
  To identify the tumor biomarkers that can best predict response to panitumumab

CONTACTS AND LOCATIONS:
Overall Officials: Michele Ghielmini, Prof, Study Chair — Oncology Institute of Southern Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siano M, Molinari F, Martin V, Mach N, Fruh M, Freguia S, Corradino I, Ghielmini M, Frattini M, Espeli V. Multicenter Phase II Study of Panitumumab in Platinum Pretreated, Advanced Head and Neck Squamous Cell Cancer. Oncologist. 2017 Jul;22(7):782-e70. doi: 10.1634/theoncologist.2017-0069. Epub 2017 Jun 7. PMID 28592616